CLINICAL TRIAL: NCT05886881
Title: Air Optix Extended Wear Contact Lenses
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLJ241-N002
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Refractive Errors
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Air Optix Aqua Sphere: Lotrafilcon B spherical soft contact lenses worn in both eyes on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Lotrafilcon B spherical soft contact lenses
- Air Optix plus HydraGlyde Sphere: Lotrafilcon B multifocal soft contact lenses with comfort additive worn in both eyes on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Lotrafilcon B spherical soft contact lenses with comfort additive
- Air Optix plus HydraGlyde Toric: Lotrafilcon B toric soft contact lenses with comfort additive worn in both eyes on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Lotrafilcon B toric soft contact lenses with comfort additive
- Biofinity Sphere: Comfilcon A spherical soft contact lenses worn in both eyes on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Comfilcon A spherical soft contact lenses
- Biofinity Toric: Comfilcon A toric soft contact lenses worn in both eyes on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Comfilcon A toric soft contact lenses

INTERVENTIONS:
Device: Lotrafilcon B spherical soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Air Optix® Aqua Sphere
  Groups: Air Optix Aqua Sphere
Device: Lotrafilcon B spherical soft contact lenses with comfort additive — Commercially available silicone hydrogel contact lenses
  Other Names: Air Optix® plus HydraGlyde® Sphere
  Groups: Air Optix plus HydraGlyde Sphere
Device: Lotrafilcon B toric soft contact lenses with comfort additive — Commercially available silicone hydrogel contact lenses
  Other Names: Air Optix® plus HydraGlyde® Toric
  Groups: Air Optix plus HydraGlyde Toric
Device: Comfilcon A spherical soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Biofinity Sphere
  Groups: Biofinity Sphere
Device: Comfilcon A toric soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Biofinity Toric
  Groups: Biofinity Toric

SUMMARY:
The purpose of this Post-Market Clinical Follow-Up (PMCF) study is to assess long term performance and safety of Air Optix Aqua Sphere, Air Optix plus HydraGlyde Sphere, and Air Optix plus HydraGlyde Toric soft contact lenses in a real-world setting when worn as extended (overnight) wear.

DETAILED DESCRIPTION:
This is a non-interventional/observational study designed as a retrospective chart review. Study sites will identify charts within their existing databases in a fair and consistent manner, e.g., reviewing all eligible charts in reverse chronological order by year of baseline visit. Subjects/charts meeting the eligibility criteria will be enrolled in the study. The data collection period is defined as any approximately 1-year to 3-year timeframe since the respective lens brand was prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Manifest refraction cylinder less than or equal to 0.75 diopter (D) in each eye at baseline (sphere wearers only);
* Best corrected visual acuity (BCVA) of 20/25 Snellen or better in each eye at baseline;
* Must have worn or be wearing Air Optix Aqua Sphere, Air Optix plus HydraGlyde Sphere, Air Optix plus HydraGlyde Toric, Biofinity Sphere or Biofinity Toric for at least 3 years in an extended wear modality, as determined by the Investigator;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any recurrent history or active anterior segment infection, inflammation or abnormality contraindicating regular contact lens wear at baseline;
* Use of systemic or ocular medications contraindicating regular contact lens wear at baseline and/or during the period of the retrospective chart collection;
* Slit lamp findings, including signs of pathological dry eye, that would contraindicate regular contact lens wear;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity (VA) with study lenses at Year 1 | Year 1
  The subject's chart will be reviewed for distance visual acuity at Year 1, defined as a visit which occurred 1 year (-2/+4 months) since baseline during which period the subject was wearing either the study or comparator lenses and a contact lens examination was performed. The Baseline visit is defined as the first office visit where an eye care practitioner provided an in-person office biomicroscopy exam to the patient before or during which a contact lens prescription for the study or comparator contact lens (lotrafilcon B or comfilcon A) was released.
Distance visual acuity (VA) with study lenses at Year 3 | Year 3
  The subject's chart will be reviewed for distance visual acuity at Year 3, defined as a visit which occurred 3 years (-2/+8 months) since baseline during which period the subject was wearing the protocol required contact lenses and a contact lens examination was performed.
Incidence of corneal infiltrative events | Up to Year 3
  The subject's chart will be reviewed for incidences of corneal infiltrative events occurring after the baseline exam.
Incidence of microbial keratitis | Up to Year 3
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Vision Health Institute, Orlando, Florida
  - Complete Eye Care of Medina, Medina, Minnesota
  - Koetting Associates, St Louis, Missouri
  - Smith Bowman Ophthalmology, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No